CLINICAL TRIAL: NCT01974479
Title: Pilot Study of Redirected Haploidentical Natural Killer Cell Infusions for B-Lineage Acute Lymphoblastic Leukemia
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended for an interim review of (CAR) CD19 research strategy for the treatment of CD19 positive ALL.
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Dr. Tan Poh Lin, Clinical Director and Senior Consultant of Paediatric Blood and Marrow Transplantation, National University Health System, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKCARCD19
Record Dates: First submitted 2013-10-20; First posted 2013-11-01 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Redirected Natural Killer Cells; Haploidentical Cell Therapy
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Intervention Model Description: To determine the feasibility, safety and efficacy of anti-CD19 redirected NK cells infusion in research participants with B-Lineage Acute Lymphoblastic Leukemia (B-ALL) who have persistent disease as determined by MRD methods after intensive chemotherapy.
Oversight: Data Monitoring Committee: No

ARMS (1):
- anti-CD19 redirected NK cells (Experimental): This is a single arm study. Intravenous Infusion of activated NK cells bearing anti-CD19-BB-zeta receptors at cell dose of 0.5 - 5 x 10^7 CD56+ cells/kg, and up to 1 x 10^8 CD56+ cells/Kg
  Interventions: Biological: anti-CD19 redirected NK cells

INTERVENTIONS:
Biological: anti-CD19 redirected NK cells — Haploidentical donor NK cells will be expanded and electroporated over 10 days and infused. NK cells will be infused at single dose on day 0. The patient will receive cyclophosphamide 60mg/kg on day - 7 , and Fludarabine 25 mg/m2/day will be given on day -6 to day -2 prior to the NK cell infusion. IL- 2 will be given subcutaneously for 6 doses every alternate day starting on day -1, for NK cell survival.
  Other Names: NKCARCD19

SUMMARY:
Modern therapy for patients with B-lineage acute lymphoblastic leukemia (ALL) is based on intensive administration of multiple drugs. In patients with relapsed disease, treatment response is generally poor; for most patients, particularly those who relapse while still receiving frontline therapy, the only therapeutic option is hematopoietic stem cell transplantation (HSCT). There is no proven curative therapy for patients who relapse after transplant.

Natural killer (NK) cells have powerful anti-leukemia activity. In patients undergoing allogeneic HSCT, several studies have demonstrated NK-mediated anti-leukemic activity. NK cell infusions in patients with leukemia have been shown to be well tolerated and void of graft-versus-host disease (GVHD) effects.

NK cell cytotoxicity is most powerful against acute myeloid leukemia (AML) cells, whereas their capacity to lyse ALL cells is generally low. We have developed a novel method to expand and redirect NK cells towards CD19, a molecule highly expressed on the surface of B-lineage ALL cells but not expressed on normal cells other than B-lymphocytes. In this method, donor NK cells are first expanded by co-culture with the cell line K562-mb15-41BBL and interleukin (IL)-2. Then, the expanded NK cells are transduced with a signaling receptor that binds to CD19 (anti-CD19-BB-zeta). NK cells expressing these receptors showed powerful anti-leukemic activity against CD19+ ALL cells in vitro and in an animal model of leukemia.

This study will assess the feasibility, safety and efficacy of infusing expanded, activated redirected NK cells into research participants with B-lineage ALL who have persistent disease after intensive chemotherapy . In this same cohort, we will study the in vivo lifespan and phenotype of these redirected NK cells.

DETAILED DESCRIPTION:
1.0. Rationale

In contrast to the well-established cytotoxicity of NK cells against AML cells, their capacity to lyse ALL cells is generally low and difficult to predict. We sought to overcome this intrinsic resistance by transducing CD56+ CD3- NK cells with chimeric receptors directed against CD19, a molecule widely expressed by malignant B cells. Expression of anti-CD19 receptors linked to CD3zeta overcame NK resistance and markedly enhanced NK cell-mediated killing of leukemic cells. This result was significantly improved by adding the 4-1BB costimulatory molecule to the chimeric anti-CD19-CD3zeta receptor: the cytotoxicity produced by NK cells expressing this construct uniformly exceeded that of NK cells whose signaling receptors lacked 4-1BB, even when natural cytotoxicity was apparent (Imai et al., Blood 2005). NK cells expressing anti-CD19 receptors also exerted vigorous anti-ALL activity in a murine model of leukemia (Shimasaki et al., Cytotherapy 2012). Our findings indicate that enforced expression of signaling receptors by NK cells might circumvent inhibitory signals, providing a novel means to enhance the effectiveness of anti-ALL NK cell therapy.

The great anti-leukemic efficacy of genetically modified NK cells shown in our preclinical studies, together with the demonstrated feasibility of infusing durable haploidentical NK cells in a non-HSCT setting and the established expertise by the NUH team in cell therapy (the only center in Asia accredited by Foundation for the Accreditation of Cellular Therapy, FACT), form a compelling rationale for the clinical testing of these NK cells.

The preparation of the key reagent (anti-CD19-BB-zeta mRNA) is finalized in the Tissue Engineering & Cell Therapy (TECT) Laboratory at NUH, where the GMP-compliant MaxCyte electroporator is located. The feasibility of large-scale expansion of NK cells has been demonstrated (Shimasaki et al. Cytotherapy 2012), and the feasibility of large-scale electroporation validated in the TECT laboratory.

We will use flow cytometric and MRD technologies, to determine the presence of persistent disease , and will include in this study only patients with a limited amount of residual disease (<1% leukemic lymphoblasts among normal bone marrow cells). We will use the same MRD methods to monitor the effects of treatment infusions. We do not expect that the conditioning regimen will have much effect by itself on leukemic cell counts, as the patients eligible for the study will have disease that is resistant to many anti-leukemic drugs. Nevertheless, because the conditioning regimen itself may have some salutary effects, it will be important to screen the peripheral blood and/or bone marrow for the presence of leukemic blast cells through all stages of the procedure, i.e., before, during, and after conditioning and after the NK cell infusion. The presence of leukemic cells in will be closely monitored by flow cytometry or PCR amplification of antigen-receptor genes (sensitivity for either method: 1 leukemic cell in 10,000) to shed some light on the relative effect of each intervention.

2.0. Hypothesis and Objectives

The main hypothesis to be tested in this study is that infusion of NK cells expressing anti-CD19-BB-zeta receptors by electroporation can produce measurable clinical responses in patients with resistant B-lineage ALL.

3.0. Primary Objectives

* To determine the feasibility and safety of redirecting NK cells with an anti-CD19 chimeric antigen receptor by mRNA electroporation in a clinical setting.
* To determine the efficacy of anti-CD19 redirected NK cells in research participants with B-lineage ALL who have persistent disease as determined by MRD methods after intensive chemotherapy.

4.0. Secondary Objectives

* To study the persistence and phenotype of redirected NK cells in research participants with B-lineage ALL who have residual disease after intensive chemotherapy.

5.0. Endpoints

In this study, treatment response will be measured by comparing MRD levels before and at several intervals after NK cell infusion.Achievement of MRD negativity in bone marrow, i.e., < 0.01% blasts by flow cytometry or PCR, will be regarded as a complete response. Partial response will be defined as ≥ 1 log decrease in MRD levels, while < 1 log decrease in MRD levels will be regarded as a no response.

Based on previous studies, donor NK cells will be eliminated in most cases by the resurgent cellular immunity of the haploidentical recipient after the effects of the transient immunosuppression caused by the conditioning regimen have ceased (typically within 1 month of infusion). Conceivably, however, NK cell engraftment may persist for a longer period with the possible risk of prolonged pancytopenia owing to NK cell killing on normal hematopoietic cells. Because of this possibility, we will plan for HSCT rescue in patients receiving redirected NK cell infusions. Indeed, for most of the patients eligible for this study, HSCT would be the treatment intervention regardless of whether they receive NK cell infusions or not. Because of these considerations, the potential benefits of NK cell therapy should outweigh its risks for those patients eligible for this study, i.e., patients with persistent leukemia for whom no other proven effective treatment is available.

Because CD19 is universally expressed on B cells including early B cell precursors, normal recipient B cell will also be a target for the donor NK cells transduced with the anti-CD19 chimeric receptors. Therefore, transient B-cell lymphopenia and hypogammaglobinemia are expected. We will monitor the CD19+ blood cell count and measure the Ig levels once a month and will give the participants intravenous immunoglobulins (IVIG) if their IgG level is lower than age-specific ranges.

6.0. Summary of Study Design

Peripheral blood cell will be collected by apheresis from donors. After ex vivo expansion for 10 days by coculture with irradiated K562-mb15-41BBL cells (Fujisaki et al, Cancer Res 2009; Lapteva et al. Cytotherapy 2012) and T-cell depletion, haploidentical NK cells will be electroporated with anti-CD19-BB-zeta mRNA. Before infusion, patients will receive immunosuppressive therapy to promote temporary engraftment of NK cells. After infusion, they will receive IL-2 to support NK cell viability and expansion in vivo. The effects of NK cell infusion will be determine by comparing MRD levels before and after treatment.

Receptor expression after electroporation is transient and typically declines after 48 hours becoming undetectable after 96 hours. Because the aim of NK cell therapy is not to induce durable immunity but to rapidly reduce tumor cell burden, and the infused NK cells are rejected by the host immune system after approximately 2 weeks of infusion, the transient nature of the expression should not significantly affect anti-tumor potential. Moreover, by using this strategy, safety concerns regarding insertional mutagenesis and long-term persistence of transduced residual T cells do not apply. In any case, we will minimize the number of residual T cells in the final product as much as possible by depleting the expanded product of T cells by using the CliniMACS device, and by limiting the number of T cells in the graft to <0.05 x 10^6/kg.

ELIGIBILITY:
Inclusion Criteria:

* NK cell RECIPIENT:

  1. Age: 0 months to 80 years old.
  2. Patients with B-lineage ALL who have persistent disease (0.01% to less than 1% as determined by flow cytometric or molecular measurements of residual disease) despite intensive standard chemotherapy .
  3. Shortening fraction greater than or equal to 25%.
  4. Glomerular filtration rate greater than or equal to 50 ml/min/1.73 m2.
  5. Pulse oximetry greater than or equal to 92% on room air.
  6. Direct bilirubin less than or equal to 3.0 mg/dL (50 mmol/L).
  7. Alanine aminotransferase (ALT) is no more than 2 times the upper limit of normal.
  8. Aspartate transaminases (AST)is no more than 2 times the upper limit of normal.
  9. Karnofsky or Lansky performance score of greater than or equal to 50.
  10. No known allergy to murine products or HAMA testing results within normal limits.
  11. No prior receipt of a gene-transfer agent (e.g. retroviral,adenoviral, lentiviral vector).
  12. Does not have a current pleural or pericardial effusion.
  13. Has a suitable adult family member donor available for NK cell donation.
  14. Has recovered from all acute NCI Common Toxicity Criteria grade II-IV non-hematologic acute toxicities resulting from prior therapy per the judgment of the PI.
  15. At least two weeks since receipt of any biological therapy, systemic chemotherapy, and/or radiation therapy.
  16. Is not receiving more than the equivalent of prednisone 10 mg daily.
  17. Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
  18. Not lactating.
* NK cell DONOR:

  1. First and second relative acceptable.
  2. 18 years of age or above.
  3. Not lactating.
  4. Greater than or equal to 3 of 6 HLA match to recipient.
  5. Meets eligibility and suitability criteria for hematopoietic cells donation as per institutional guidelines.
  6. Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).

Exclusion Criteria:

* Failure to meet any of the inclusion criteria.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Disease Response Criteria - Minimal Disease Residual (MRD) Monitoring | 1 Month Post NK Cell Infusion
  Treatment response will be measured by comparing MRD levels before and 1 month after NK cell infusion. Achievement of MRD negativity in bone marrow, i.e., < 0.01% blasts by flow cytometry or PCR, will be regarded as a complete response. Partial response will be defined as ≥ 1 log decrease in MRD levels, while < 1 log decrease in MRD levels will be regarded as no response.

CONTACTS AND LOCATIONS:
Overall Officials: Poh Lin Tan, Principal Investigator — NUHS Singapore; Dario Campana, Principal Investigator — NUHS Singapore
Locations (1):
- Department of Paediatrics, National University Health System, Singapore, Singapore

REFERENCES:
- [Background] Imai C, Iwamoto S, Campana D. Genetic modification of primary natural killer cells overcomes inhibitory signals and induces specific killing of leukemic cells. Blood. 2005 Jul 1;106(1):376-83. doi: 10.1182/blood-2004-12-4797. Epub 2005 Mar 8. PMID 15755898
- [Background] Shimasaki N, Fujisaki H, Cho D, Masselli M, Lockey T, Eldridge P, Leung W, Campana D. A clinically adaptable method to enhance the cytotoxicity of natural killer cells against B-cell malignancies. Cytotherapy. 2012 Aug;14(7):830-40. doi: 10.3109/14653249.2012.671519. Epub 2012 Mar 29. PMID 22458956
- [Background] Fujisaki H, Kakuda H, Shimasaki N, Imai C, Ma J, Lockey T, Eldridge P, Leung WH, Campana D. Expansion of highly cytotoxic human natural killer cells for cancer cell therapy. Cancer Res. 2009 May 1;69(9):4010-7. doi: 10.1158/0008-5472.CAN-08-3712. Epub 2009 Apr 21. PMID 19383914
- [Background] Lapteva N, Durett AG, Sun J, Rollins LA, Huye LL, Fang J, Dandekar V, Mei Z, Jackson K, Vera J, Ando J, Ngo MC, Coustan-Smith E, Campana D, Szmania S, Garg T, Moreno-Bost A, Vanrhee F, Gee AP, Rooney CM. Large-scale ex vivo expansion and characterization of natural killer cells for clinical applications. Cytotherapy. 2012 Oct;14(9):1131-43. doi: 10.3109/14653249.2012.700767. Epub 2012 Aug 17. PMID 22900959
- [Derived] Del Zotto G, Marcenaro E, Vacca P, Sivori S, Pende D, Della Chiesa M, Moretta F, Ingegnere T, Mingari MC, Moretta A, Moretta L. Markers and function of human NK cells in normal and pathological conditions. Cytometry B Clin Cytom. 2017 Mar;92(2):100-114. doi: 10.1002/cyto.b.21508. Epub 2017 Feb 12. PMID 28054442